CLINICAL TRIAL: NCT05118503
Title: Personalized Patient and Caregiver Education After Stroke
Acronym: MyStroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Christopher Favilla, Assistant Professor of Neurology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 833723
Record Dates: First submitted 2021-10-12; First posted 2021-11-12 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Stroke, Acute; Stroke, Ischemic; Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized education app (Active Comparator): A customized URL-based platform will present brief education videos addressing a patients stroke etiology, risk factors, stroke prevention medications, and post-stroke lifestyle issues. This URL will be made available to the patient and caregiver.
  Interventions: Behavioral: Customized education
- Standard of care discharge education (Placebo Comparator): Standard discharge education is performed by the bedside nurse at the time of hospital discharge.
  Interventions: Behavioral: Standard of care discharge education

INTERVENTIONS:
Behavioral: Customized education — Half of subjects will receive access to a customized app that will include brief educational videos that have been selected for each patient based on their medical history. These videos will address stroke etiology, underlying risk factors, and stroke prevention medications.
  Arms: Customized education app
Behavioral: Standard of care discharge education — Half of subjects will be randomized to receive typical discharge education, per the institutional guidelines for standard of care education for stroke patients.
  Arms: Standard of care discharge education

SUMMARY:
This is a randomized pilot trial to evaluate the impact of a customizable stroke education app (vs standard of care discharge education) on patient satisfaction and education retention. The impact of the intervention will be assessed 7, 30, and 90 days post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for ischemic stroke
* At least 18 years old
* Patient or caregiver has access to a smart phone, tablet or computer
* Being discharged to either home or acute rehab

Exclusion Criteria:

* Patient or caregivers unable or unwilling to access the customized app with a smartphone, tablet, or computer
* Being discharged to a skilled nursing facility
* moderate-to-severe aphasia at the time of enrollment (as per NIHSS scoring) if patient is being enrolled without a caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction survey | Day 90
  Likert-style survey assessing patient satisfaction and perception of the stroke education they received.
Stroke etiology awareness | Day 90
  accurate knowledge of stroke etiology (0=incorrect; 1=correct)
Stroke Patient Education Retention (SPER) survey | Day 90
  Validated measure of stroke patient education as it pertains to their stroke etiology and risk factors with scores of 0-10
EuroQOL-VAS | Day 90
  validated quality of life metric, with scores of 0-100

SECONDARY OUTCOMES:
Stroke etiology awareness | Day 7
  accurate knowledge of stroke etiology (0=incorrect; 1=correct)
Stroke etiology awareness | Day 30
  accurate knowledge of stroke etiology (0=incorrect; 1=correct)
Stroke risk factor awareness. 7 days | Day 7
  accurate knowledge of stroke risk factors (0=incorrect; 1=correct)
Stroke risk factor awareness, 30 days | Day 30
  accurate knowledge of stroke risk factors (0=incorrect; 1=correct)
Stroke risk factor awareness, 90 days | Day 90
  accurate knowledge of stroke risk factors (0=incorrect; 1=correct)
Stroke prevention med awareness, 7 days | Day 7
  accurate knowledge of stroke prevention medications (0=incorrect; 1=correct)
Stroke prevention med awareness, 30 days | Day 30
  accurate knowledge of stroke prevention medications (0=incorrect; 1=correct)
Stroke prevention med awareness, 90 days | Day 90
  accurate knowledge of stroke prevention medications (0=incorrect; 1=correct)
Patient satisfaction, 7 days | Day 7
  Likert-style survey assessing patient satisfaction and perception of the stroke education
Patient satisfaction, 30 days | Day 30
  Likert-style survey assessing patient satisfaction and perception of the stroke education
SPER, 7 days | Day 7
  Stroke Patient Education Retention (SPER) survey
SPER, 30 days | Day 30
  Stroke Patient Education Retention (SPER) survey

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Favilla, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Favilla CG, Reehal N, Cummings SR, Burdett R, Stein LA, Shakibajahromi B, Yuan K, Sloane KL, Kasner SE. Personalized Video-Based Educational Platform to Improve Stroke Knowledge: A Randomized Clinical Trial. J Am Heart Assoc. 2024 Aug 6;13(15):e035176. doi: 10.1161/JAHA.124.035176. Epub 2024 Jul 31. PMID 39082426